CLINICAL TRIAL: NCT02947048
Title: A Randomized, Placebo-controlled Phase 2 Study With Open-Label and Double-Blind Portions to Evaluate the Safety of L1-79 in Adolescent and Young Adult Males With Autism
Brief Title: Safety of L1-79 in Adolescent and Adult Males With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yamo Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT 02-121
Record Dates: First submitted 2016-05-25; First posted 2016-10-27 (Estimated); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 100 mg open (Experimental): open-label lead-in 100 mg L1-79 t.i.d.
  Interventions: Drug: L1-79
- 100 mg blinded (Experimental): blinded and randomized 100 mg L1-79 t.i.d.
  Interventions: Drug: L1-79
- 200 mg open (Experimental): open-label lead-in 200 mg L1-79 t.i.d.
  Interventions: Drug: L1-79
- 200 mg blinded (Experimental): blinded and randomized 200 mg L1-79 t.i.d.
  Interventions: Drug: L1-79
- Placebo (Placebo Comparator): placebo t.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L1-79
  Other Names: D,L-α-Methyltyrosine
  Arms: 100 mg blinded; 100 mg open; 200 mg blinded; 200 mg open
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a five-arm designed to assess the safety of L1-79 that incorporates 15 prospectively randomized, placebo controlled patients and 5 open label patients at either 100 tid (three times daily) or 200 tid dosing for 28 days. The open label patients will be assessed for the purpose of understanding PK/PD and to determine if there are any EKG changes associated with the administration of L1-79. Additional safety information will be provided by the 30 patients randomized 2:1 active:placebo.

DETAILED DESCRIPTION:
Protocol Number: HT 02-121

Protocol Title: Phase 2 Safety Study of L1-79 for the Treatment of Autism Study Phase: 2

The first cohort of 20 patients to be enrolled will all receive L1-79 100 mg t.i.d., and will be comprised of 3 groups of patients. The first group of patients to receive 100 mg will differ from the others in that they will get blood samples drawn for PK analysis and EKGs will be taken. The safety and PK data from this group will be submitted for FDA review and acceptance before the 200 mg t.i.d. cohort will be enrolled. The remaining 15 patients in this cohort will be randomized to receive either L1-79 100 mg t.i.d. or placebo on a 2:1 basis (2 L1-79 patients for each placebo patient). While the FDA is reviewing the data from the first 5 patients all 100 mg t.i.d. patients will continue to be treated.

The second cohort is identical to the first. The initial 5 patients to be enrolled will differ from the others in that they will get blood samples drawn for PK analysis and EKGs will be taken. The remaining 15 patients in this cohort will be randomized to receive either L1-79 200 mg t.i.d. or placebo on a 2:1 active:placebo.

Sample Size: N=40

* Group 1 (n=5) open100mg L1-79 (1x100mg capsule+1 placebo capsule)
* Group 2 (n=10) blind100mg L1-79 (1x100mg capsule+1 placebo capsule)
* Group 3 (n=5) open200 mg L1-79 (2x100 mg capsules)
* Group 4 (n=10) blind200 mg L1-79 (2x100 mg capsules)
* Group 5 (n=10) Placebo (2 placebo capsules) All Groups will receive the assigned study drug three-times daily

Study Population: Male subjects with autism between the ages of 13 and 21 years of age who meet the entry criteria and who are able to complete standardized measures allowing them to participate in this study.

Evaluation Schedule: Subjects will be evaluated within one week prior to study accession, and weekly throughout the dosing period, and again 4 weeks after the cessation of treatment. The Assigned Dosage Groups (Groups 1 and 3) will have PK blood draws and EKG the randomized group will not have.

Safety Measures: All Groups will have regularly scheduled complete history and physical examination that includes orthostatic blood pressure measurements, vital signs, CBC, differential, platelet counts, urine analysis, and serum analytes including: total protein, albumin, glucose, BUN, creatinine, direct and total bilirubin, alkaline phosphatase, phosphorous, calcium, AST, ALT, sodium, potassium, chloride, bicarbonate, T4, TSH, and adverse events assessments. The Assigned Groups (1 and 3) will also have electrocardiograms taken at the study screening visit and weekly throughout the treatment interval.

ELIGIBILITY:
Inclusion Criteria:

1. Males who are not sexually active
2. 12 and 21 years of age
3. Signed informed consent
4. Normal clinical laboratory values
5. DSM-5 compliant diagnosis of autism spectrum disorder, confirmed by the Autistic Diagnosis Interview Review (ADIR), and by the Autism Diagnosis Observation Schedule (ADOS) score consistent with a diagnosis of autism
6. No more than one concomitant medication for the treatment of autism, on a stable for at least 2 weeks prior to enrollment and no planned changes in psychosocial interventions during the trial
7. No medications for any other pathology

Exclusion Criteria:

1. Any co-morbidities, including Fragile-X syndrome, epilepsy, Retts syndrome, ADHD, or other disease or syndrome aside from autism that requires treatment
2. Any other psychiatric disorder, or out of range lab values
3. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, alcohol use disorder
4. Active medical problems: unstable seizures (>2 in past month)
5. Concomitant physical illness

Ages: 12 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rothman, PhD, Study Director — Yamo Pharmaceuticals
Locations (2):
- United States (2):
  - Eric Bartky MD, Bartky Health Care Center, Livingston, New Jersey
  - F. Peter Halas MD, Sea Girt Pediatrics, Sea Girt, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg Open: open-label lead-in L1-79 100 mg tid
- 100 mg Blinded: blinded and randomized L1-79 100 mg tid
- Placebo (100 mg Cohort); Placebo (200 mg Cohort): blinded and randomized placebo tid
- 200 mg Open: open-label lead-in L1-79 200 mg tid
- 200 mg Blinded: blinded and randomized L1-79 200 mg tid
Period: Overall Study
Arm/Group | 100 mg Open | 100 mg Blinded | Placebo (100 mg Cohort) | 200 mg Open | 200 mg Blinded | Placebo (200 mg Cohort)
Started | 5 | 10 | 5 | 6 | 11 | 5
Safety Population (For safety analyses both placebo groups were combined.) | 5 | 10 | 5 | 6 | 11 | 5
Efficacy Population (The efficacy population includes patients enrolled in the double-blind portion of the study. Two patients were omitted for the efficacy population in Cohort 1 (1 patient in placebo and 1 patient in L1-79 100 mg TID group) because there was apparent confusion in the assigned-vs.-received drug kit numbers. These patients were included in the safety population.) | 0 | 9 | 4 | 0 | 11 | 5
Completed | 5 | 10 | 5 | 5 | 10 | 4
Not Completed | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- 100 mg Open: open-label lead-in 100 mg L1-79 t.i.d.
  L1-79
- 100 mg Blinded: blinded and randomized 100 mg L1-79 t.i.d.
  L1-79
- Placebo Blinded (100 mg Cohort): blinded and randomized placebo t.i.d.
  Placebo (100 mg cohort)
- 200 mg Open: open-label lead-in 200 mg L1-79 t.i.d.
  L1-79
- 200 mg Blinded: blinded and randomized 200 mg L1-79 t.i.d.
  L1-79
- Placebo Blinded (200 mg Cohort): blinded and randomized placebo t.i.d.
  Placebo (200 mg cohort)
- Total: Total of all reporting groups
Arm/Group | 100 mg Open | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Open | 200 mg Blinded | Placebo Blinded (200 mg Cohort) | Total
Number analyzed (Participants) | 5 | 10 | 5 | 6 | 11 | 5 | 42
Age, Continuous [Mean (Full Range); unit: years] | 16.2 [13 to 19] | 16.1 [13 to 20] | 15.3 [13 to 17] | 15.8 [13 to 18] | 16.4 [12 to 20] | 16.6 [12 to 19] | 16.1 [12 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 10 | 5 | 6 | 11 | 5 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 0 | 3
  White | 4 | 10 | 2 | 5 | 9 | 5 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 5 | 6 | 11 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of Participants with On-treatment Adverse Events.
  To be conservative, it was pre-specified that all placebo data be combined (open-label, first cohort, and second cohort) for the safety population. For the efficacy population open-label data was excluded due to potential bias and placebo arms from the first and second cohort were presented separately due to differences in efficacy questionnaires completion in the first and second cohorts. Theses differences were not relevant to the adverse event data.
Time Frame: 4 weeks
Population: Safety Population. Note that all Placebo data (open-label, first cohort and second cohort) is combined for the safety population. However for the efficacy population the open-label data is excluded and placebo arms from the first cohort and second cohort are presented separately because in the first cohort questionnaires were filled out at home by patients and in the second cohort they were completed in clinic with study staff.
Measure: Number; unit: participants
Groups:
- 100 mg Open: open-label lead-in 100 mg L1-79 tid
- 100 mg Blinded: blinded and randomized 100 mg L1-79 tid
- 200 mg Open: open-label lead-in 200 mg L1-79 tid
- 200 mg Blinded: blinded and randomized 200 mg L1-79 tid
- Placebo Blinded (100 mg Cohort): blinded and randomized placebo tid (100 mg cohort)
- Placebo Blinded (200 mg Cohort): blinded and randomized placebo tid (200 mg cohort)
Arm/Group | 100 mg Open | 100 mg Blinded | 200 mg Open | 200 mg Blinded | Placebo Blinded (100 mg Cohort) | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 5 | 10 | 6 | 11 | 5 | 5
participants
  any adverse event | 2 | 1 | 2 | 6 | 5 | 5
  diarrhea | 0 | 0 | 0 | 3 | 0 | 0
  fatigue | 0 | 0 | 1 | 0 | 0 | 0
  pyrexia | 0 | 0 | 1 | 0 | 0 | 0
  seasonal allergy | 0 | 0 | 1 | 0 | 0 | 0
  ear infection | 0 | 0 | 0 | 1 | 0 | 0
  nasopharyngitis | 0 | 0 | 0 | 0 | 0 | 1
  otitis externa | 0 | 0 | 0 | 1 | 0 | 0
  amylase increased | 0 | 0 | 0 | 0 | 0 | 1
  blood thyroid stimulating hormone increased | 0 | 0 | 0 | 1 | 0 | 0
  crystal urine present | 0 | 0 | 0 | 2 | 0 | 0
  generalized tonic-clonic seizure | 0 | 0 | 0 | 1 | 0 | 0
  syncope | 0 | 1 | 0 | 0 | 0 | 0
  agitation | 0 | 0 | 0 | 0 | 0 | 1
  anxiety | 1 | 0 | 0 | 1 | 0 | 0
  confusional state | 1 | 0 | 0 | 0 | 0 | 0
  intentional self-injury | 2 | 0 | 0 | 0 | 0 | 1
  irritability | 2 | 0 | 0 | 0 | 0 | 0
  urinary incontinence | 0 | 0 | 0 | 0 | 0 | 1
  cough | 0 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale (CGI)
Description: The Clinical Global Impression (CGI) has two components: the CGI-Severity (CGI-S), which rates illness severity, and the CGI-Improvement (CGI-I), which rates the change in illness severity from baseline.
  The CGI-S is rated on the following seven-point scale with 1 being normal and 7 being among the most extremely ill subjects. The CGI-I score is rated on a seven-point scale with 1 being very much improved and 7 being very much worse.
  Higher values of the CGI-S score indicate a "worse" state. CGI-I scores of 5 or greater indicate decline, CGI I scores of 3 or lower indicate improvement, and a CGI-I score of 4 indicates no change.
Time Frame: Week 0 and Week 4
Population: Efficacy Population Note that for the efficacy population open-label data is excluded and placebo arms from the first cohort and second cohort are presented separately because in the first cohort questionnaires were filled out at home by patients and in the second cohort they were completed in clinic with study staff.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 9 | 4 | 10 | 4
score on a scale
  Change from Baseline in Clinical Global Impression - Severity | -0.5 (0.2) | -0.2 (0.3) | -0.8 (0.3) | -0.3 (0.4)
  Clinical Global Impression - Improvement | 3.0 (0.3) | 2.8 (0.4) | 2.8 (0.2) | 2.8 (0.4)
Statistical Analysis 1: Comparison: 100 mg Blinded vs Placebo Blinded (100 mg Cohort); Clinical Global Impression - Severity; Test type: Superiority; p = 0.61, ANCOVA; Mean Difference (Final Values) = -0.22, Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: 200 mg Blinded vs Placebo Blinded (200 mg Cohort); Clinical Global Impression - Severity; Test type: Superiority; p = 0.33, ANCOVA; Mean Difference (Final Values) = -0.53, Standard Error of Mean 0.52
Statistical Analysis 3: Comparison: 100 mg Blinded vs Placebo Blinded (100 mg Cohort); Clinical Global Impression - Improvement; Test type: Superiority; p = 0.61, ANCOVA; Mean Difference (Final Values) = 0.25, Standard Error of Mean 0.47
Statistical Analysis 4: Comparison: 200 mg Blinded vs Placebo Blinded (200 mg Cohort); Clinical Global Impression - Improvement; Test type: Superiority; p = 0.91, ANCOVA; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.43

3. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scale - 2nd Edition Socialization Standard Score
Description: The Vineland Adaptive Behavior Scales, Second Edition (VABS-II) indicates adaptive functioning and consists of four major domains. Only the communication and socialization domains were done in this study. The VABS-II data is comprised of Socialization.
  Socialization Standard Scores may range from 20 to 160, with a population mean of 100 and a standard deviation of 15. Lower Vineland Adaptive Behavior Socialization Standard Scores indicate a "worse" state. A positive value of change from baseline indicates improvement.
Time Frame: Day 0 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 5 | 2 | 7 | 2
score on a scale | -4.2 (12.1) | 0.0 (0.0) | 7.6 (11.9) | 1.5 (2.1)

4. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scale - 2nd Edition Communication Standard Score
Description: The Vineland Adaptive Behavior Scales, Second Edition (VABS-II) indicates adaptive functioning and consists of four major domains. Only the communication and socialization domains were done in this study. The VABS-II is comprised of Communication.
  Communication Standard Scores may range from 20 to 160, with a population mean of 100 and a standard deviation of 15. Lower Vineland Adaptive Behavior Communication Standard Scores indicate a "worse" state. A positive value of change from baseline indicates improvement.
Time Frame: Week 0 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 8 | 3 | 7 | 2
score on a scale | 10.1 (16.6) | 7.7 (10.8) | 2.7 (4.3) | 3.0 (2.8)

5. Secondary Outcome: Change From Baseline in the Autism Diagnostic Observation Schedule 2nd Edition (ADOS-2) Overall Total Score
Description: The Autism Diagnostic Observation Schedule 2nd Edition (ADOS-2) is the "Gold Standard" for assessing severity of ASD and position on the autism spectrum. The ADOS-2 is a semi-structured, standardized assessment of: Communication, Social interaction, Play, and Restricted and repetitive behaviors. The total scores range from 15 to 60, and the cut-off score to determine autism is 30. More specifically, a score of <30 is classified as non-autism, a score of 30-36 is classified as mild to moderate autism, and a score of ≥37 is classified as severe autism.
  A higher ADOS-2 value indicates a "worse" state. A negative value of change from baseline indicates an improvement.
Time Frame: Day 0 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 9 | 4 | 10 | 4
score on a scale | -0.6 (1.7) | 0.3 (1.0) | -1.0 (2.2) | -0.3 (3.0)

6. Secondary Outcome: Change From Baseline in the Social Responsiveness Scale - 2nd Edition (SRS-2) Total T-score
Description: Social Responsiveness Scale - 2nd edition (SRS-2) identifies social impairment associated with ASD and quantifies its severity. Raw and T-scores will be collected for SRS-2 Total, Social Awareness, Social Cognition, Social Communication, Social Motivation, Restricted Interest and Repetitive Behavior, DSM-5 Social Communication, and DSM-5 Restrictive Interest and Repetitive Behavior. Each domain has a varied but similar ranges of possible scores from 32 points-114 points. All T-scores have a mean of 50 points with a standard deviation of 10 points.
  A higher SRS-2 total T-score indicates greater impairment. A negative change from baseline indicates improvement.
Time Frame: Week 0 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 8 | 4 | 10 | 4
score on a scale
  total T-score | -0.4 (6.2) | -3.8 (9.6) | -8.6 (11.1) | -9.3 (9.8)
  social awareness T-score | 1.0 (11.3) | -0.8 (1.5) | -2.8 (10.3) | -8.0 (14.9)
  social cognition T-score | 0.4 (5.4) | -2.3 (5.3) | -11.4 (20.9) | -7.5 (14.1)
  social communication T-score | 1.1 (7.1) | -3.0 (9.0) | -8.9 (11.4) | -9.3 (12.6)
  social motivation T-score | -1.4 (9.2) | 0.8 (12.8) | -11.5 (12.9) | -6.8 (4.9)
  RRB T-score | -0.4 (9.3) | -9.8 (14.0) | -8.7 (13.5) | -7.3 (7.2)
  DSM-5 social communication interaction T-score | 0.6 (5.4) | -2.3 (8.9) | -8.3 (10.6) | -9.0 (11.5)
  DSM-5 RRB T-score | -0.4 (9.3) | -9.8 (14.0) | -8.7 (13.5) | -7.3 (7.2)

7. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist - Community (ABC-C)
Description: The Aberrant Behavior Checklist - Community (ABC-C) is a 58-symptom checklist for assessing problem behaviors of children and adults with developmental disabilities (intellectual disability, ASD, cerebral palsy, epilepsy) that resolve onto five subscales. The subscales and the respective number of items are as follows: (a) irritability (15 items, scores range from 0-45), (b) lethargy/social withdrawal (16 items, scores range from 0-48), (c) stereotypic behavior (7 items, scores range from 0-21), (d) hyperactivity/noncompliance (16 items, scores range from 0-48), and (e) inappropriate speech (4 items, scores range from 0-12).
  Higher ABC-C subscale scores indicates a "worse" outcome. A negative value of change from baseline indicates improvement.
Time Frame: Week 0 to Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 9 | 4 | 10 | 4
score on a scale
  irritability and agitation | -0.9 (2.0) | -5.3 (3.8) | -3.1 (6.5) | -4.5 (4.8)
  lethargy and social withdrawal | -1.6 (6.7) | -3.5 (6.8) | -5.4 (6.2) | -8.0 (4.1)
  stereotypic behavior | 1.9 (3.3) | -1.0 (2.9) | -2.0 (2.9) | -2.8 (1.7)
  hyperactivity and noncompliance | 0.4 (3.9) | -6.7 (3.1) | -4.6 (9.4) | -5.5 (6.0)
  inappropriate speech | 0.0 (1.7) | -1.3 (1.2) | -2.1 (2.6) | -2.5 (4.0)

8. Secondary Outcome: Change From Baseline in the Repetitive Behavior Scale - Revised (RBS-R) Total Score
Description: The RBS-R is a 43-item self-report questionnaire that is used to measure the breadth of repetitive behavior in children, adolescents, and adults with Autism Spectrum disorders. Behaviors are rated on a 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. The total score is the sum of all 6 subscale scores and ranges from 0-127, stereotypic behavior ranges from 0-18, self-injurious behavior ranges from 0-24, compulsive behavior ranges from 0-24, ritualistic behavior ranges from 0-18, sameness behavior ranges from 0-33 and restricted behaviors ranges from 0-12.
  A higher RBS-R score indicates a "worse" state. A negative value of change from baseline indicates an improvement.
Time Frame: Week 0 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Blinded | Placebo Blinded (100 mg Cohort) | 200 mg Blinded | Placebo Blinded (200 mg Cohort)
Number analyzed (Participants) | 9 | 3 | 10 | 4
score on a scale
  total score | -3.2 (7.8) | -9.3 (12.7) | -17.6 (24.9) | -16.5 (6.0)
  stereotypic behavior | -0.6 (1.7) | -2.3 (4.0) | -1.9 (2.9) | -0.5 (2.6)
  self-injurious behavior | -2.2 (5.3) | -2.3 (4.9) | -2.0 (4.0) | -2.3 (3.3)
  compulsive behavior | -1.2 (3.6) | -0.7 (0.6) | -3.0 (5.1) | -2.5 (1.7)
  ritualistic behavior | 0.1 (2.8) | 0.0 (0.0) | -3.4 (4.2) | -6.0 (2.6)
  sameness behavior | -0.7 (2.0) | -2.3 (3.2) | -4.6 (7.3) | -3.3 (1.5)
  restricted behavior | 1.3 (2.6) | -1.7 (1.5) | -2.7 (2.9) | -2.0 (1.6)

ADVERSE EVENTS:
Time Frame: From the time of screening to the end of the study (28-day treatment period with 4-week post-treatment follow-up)
Description: To be conservative, it was pre-specified that all placebo data be combined (open-label, first cohort, and second cohort) for the safety population. For the efficacy population open-label data was excluded due to potential bias and placebo arms from the first and second cohort were presented separately due to differences in efficacy questionnaires completion in the first and second cohorts. Theses differences were not relevant to the adverse event data.
Arm/Group | 100 mg Open | 100 mg Blinded | 200 mg Open | 200 mg Blinded | Placebo Blinded (100 mg Cohort) | Placebo Blinded (200 mg Cohort)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/6 | 0/11 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/6 | 0/11 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 1/10 | 2/6 | 6/11 | 0/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Open (N=5) | 100 mg Blinded (N=10) | 200 mg Open (N=6) | 200 mg Blinded (N=11) | Placebo Blinded (100 mg Cohort) (N=5) | Placebo Blinded (200 mg Cohort) (N=5)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ear infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
blood TSH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intentional self injury (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
irritability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study enrolled a small number of patients and was not powered to detect statistically significant changes in efficacy parameters. Also note that assessments (except CGI and ADOS-2) for 100 mg cohort were completed by caregivers at home. Due to missing/incomplete data for endpoints completed at home, study procedures changed for 200 mg cohort and assessments were completed in clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02947048/Prot_SAP_000.pdf